CLINICAL TRIAL: NCT04175314
Title: Severity of Periodontal Recession by Patient and Associated Risk Factors in France.
Brief Title: Severity of Periodontal Recession and Associated Risk Factors in France.
Acronym: Recession
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2016/RECESSION-BISSON/MS
Record Dates: First submitted 2019-08-20; First posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-07

CONDITIONS: Periodontal Recessions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case -: Patient presenting one or more periodontal recession more than 1mm of height
  Interventions: Other: Clinical examination of gingival tissues
- Control-: Patient presenting no periodontal recession or recession of less than 1 mm of height
  Interventions: Other: Clinical examination of gingival tissues

INTERVENTIONS:
Other: Clinical examination of gingival tissues — Measure of the periodontal recession

SUMMARY:
The severity of periodontal recessions for each examined patient during dental consultation was evaluated. Moreover, the description of the number of periodontal recessions in patients with good health during dental consultation, the associated risk factors and evaluation of the number of recessions which need surgical therapy were realized.

ELIGIBILITY:
Inclusion Criteria:

Case:

* patients aged from 20 to 50 years
* patients with recession of more than 1mm
* patient with good health
* patients who aggreed to participate to the study

Controls:

* patients aged from 20 to 50 years
* patients with no recession or recession less than 1mm
* patient with good health
* patients who aggreed to participate to the study

Exclusion Criteria:

* patients with periodontitis
* patients with recession of Class III and IV of modified Miller classification
* patients with previous muco-gingival surgery
* patients pregnant, breatheeding
* patients refusing to participate to the study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients are selected during a dental consultation.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2021-02-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of periodontal recession severity | Observation at day 1
  Measure of the height and the width of periodontal recession (millimeter)

SECONDARY OUTCOMES:
Number of recessions for each patient | Observation at day 1
  Evaluation of the number of recessions for each patient
Associated risk factors | Observation at day 1
  Evaluation of smoking status, general health, periodontum and dental parameters, evaluation of toothbrush and dental treatment
Number of participants with recession-related adverse events as assessed by questionnaire | Observation at day 1
  Evaluation of the needs of surgical treatment of the periodontal recessions observed according to pain evaluated by questionnaire
Frequency of periodontal recession according to the modified Miller classifcation | Observation at day 1
  Measure of the periodontal recession according to the modified Miller classification

CONTACTS AND LOCATIONS:
Overall Officials: Catherine BISSON, Principal Investigator — Central Hospital
Locations (5):
- France (5):
  - CHU Henri Mondor, Créteil
  - CHU, Montpellier
  - CHU, Nancy
  - CHU Saint Roch, Nice
  - CHU Ragueil, Toulouse